CLINICAL TRIAL: NCT04887649
Title: Randomized, Controlled, Double Blind, to Evaluate the Postpartum Analgesia With Epidural Morphine: Analgesic Effect of Two Different Doses Compared to Placebo
Acronym: IMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7245408
Record Dates: First submitted 2011-10-13; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Labor Pain
Keywords: Epidural opioid; Morphine; Postpartum pain; Analgesia; Perineorraphy
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Morphine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Patients en treatment whit placebo, salIne solution in peridural cateter
  Interventions: Drug: saline solution
- Morphine (Active Comparator): Epidural Catheter morphine 2mg
  Interventions: Drug: Morphine
- morphine (Active Comparator): Epidurla cateter morphine 3 mg
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — morphine 3 mg
  Other Names: Random code numbers
  Arms: Morphine; morphine
Drug: saline solution — 4 cc of saline solution in epidural cateter in postpartum
  Other Names: Random code numbers
  Arms: Placebo
Drug: Morphine — morphine 2 mg for epidural cateter in postpartum
  Other Names: Random code numbers
  Arms: Morphine; morphine

SUMMARY:
This study aims to assess the analgesic effect of two different doses of epidural morphine for postpartum analgesia management. Previous studies have shown that conventional management of postpartum pain (acetaminophen, NSAIDs) is insufficient, in the investigators country is wasted using the epidural catheter is placed as part of the analgesic management of pregnant women in labor.

DETAILED DESCRIPTION:
The intervention is the epidural administration of morphine in two doses 2mg and 3mg different vs placebo 1 hour after delivery care maternal vaginal in patients who received epidural analgesia in labor, in order to evaluate the analgesic effectiveness post operations of the different doses vs placebo.

In the analysis to determine whether the proposed levels are effective for postpartum pain control was carried out by determining the differences between experimental groups and control group, and in examining the statistical significance of the differences found by applying the relevant tests according to whether the variable is normally distributed or not.

The main variables analyzed were:

rating of pain intensity, number of analgesics required required dose of analgesics used to achieve adequate control pain, number of pain episodes and percentage of patients free of these episodes, duration of action of the dose used.

Similar analysis was determined by the incidence of side effects, in particular those described in classic form, pruritus, nausea and vomiting, urinary retention, and respiratory depression

Were classified into three groups: two experimental and one control group.

Experimental Group 1 will receive 10 ml of solution prepared as follows:

2 mg of morphine diluted in 0.9% normal saline

Experimental Group 2 will receive 10 ml of solution prepared as follows:

3 mg of morphine diluted in 0.9% normal saline

The control group will receive 10 ml of normal saline (SSN).

The randomization codes were kept in a sealed envelope so individual, and the envelopes were guarded and uncovered after a eligible to participate in the study agreed to be included and signed the informed consent.

Anesthesia Technique for the Study

In ASA II patients in labor who were initiates of labor analgesia with epidural catheter has been placed ideally at the level of L3-L4 (Tuohy catheter conventional number 18, introduced by loss of resistance technique) .

The patients were started a conventional dose of analgesia with bupivacaine 0.5% + fentanyl 100mcg 10mg 10cc carried in a bolus. Administered bupivacaine + 10 mg bolus of fentanyl 100mcg as needed to strengthen the epidural analgesia

or Infusion Bupivacaine 0.125% + Fentanyl 100mcg%

In a 10cc bolus then 8-16CC hours

In patients 1 hour after having her expulsive morphine were previously applied in laboratory and packaged in disregard of the anesthesiologist applied morphine 2mg - 3mg or saline placebo.

The dose will be applied 1 hour after birth in search of having no residual analgesic effect of local anesthetic and opioid epidural analgesia initially applied.

All patients will be managed with conventional analgesia performed in the institution acetaminophen 1 g every 6 hours VO

If additional merit the first choice analgesic diclofenac 75mg IM is, if no answer will apply a dose of 100mg tramadol or morphine IV in titrated only if warranted more analgesia.

For all patients will have availability of naloxone in case of respiratory depression.

Patients will be observed for 24 hours with monitoring the consumption of other analgesics, pain visual analog scale, which is evaluated at the time of the application of morphine, 2h, 4h, 6h 12h and 24h after application of morphine. Also evaluated variables such as development of pruritus, nausea, vomiting, urinary retention and assessment of respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients postpartum vaginal conventional analgesia management of your labor
* ASA II
* Do not include patients with history of allergy to morphine.
* Patients who agreed to be included in the study but did not sign informed consent.

Exclusion Criteria:

* Submit a complication that makes it difficult postoperative pain assessment or adverse effects after surgery.
* Patients who, after having been included, express their desire to be excluded. Patients with incomplete follow-up.id
* Did not include patients who have absolute contraindications for epidural anesthesia, or could not provide informed consent, as in the following cases: local infection at the site of administration, systemic infection, bleeding disorders, disease of the spine , mental patients, drug history, sleep apnea, history of headache post-puncture headache or frequent any kind.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The analgesic efficacy: : pain intensity rating | The first 24 hours after administration
  The analgesic efficacy at controlling pain after delivery

SECONDARY OUTCOMES:
the incidence of side effects | the first 24 hours after administration
  In particular those described in the literature, such as pruritus, nausea, vomiting, urinary retention and respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Dario J Perea, Medical, Study Chair — Universidad Nacional de Colombia
Locations (1):
- Universidad Nacional; Maternal and Child Institute, Bogotá, Colombia

REFERENCES:
- [Background] Wang JK, Nauss LA, Thomas JE. Pain relief by intrathecally applied morphine in man. Anesthesiology. 1979 Feb;50(2):149-51. doi: 10.1097/00000542-197902000-00013. No abstract available. PMID 373503
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Macarthur A, Imarengiaye C, Tureanu L, Downey K. A randomized, double-blind, placebo-controlled trial of epidural morphine analgesia after vaginal delivery. Anesth Analg. 2010 Jan 1;110(1):159-64. doi: 10.1213/ANE.0b013e3181c30f78. Epub 2009 Nov 12. PMID 19910627
- [Background] Goodman SR, Drachenberg AM, Johnson SA, Negron MA, Kim-Lo SH, Smiley RM. Decreased postpartum use of oral pain medication after a single dose of epidural morphine. Reg Anesth Pain Med. 2005 Mar-Apr;30(2):134-9. doi: 10.1016/j.rapm.2004.11.010. PMID 15765455
- [Background] Behar M, Magora F, Olshwang D, Davidson JT. Epidural morphine in treatment of pain. Lancet. 1979 Mar 10;1(8115):527-9. doi: 10.1016/s0140-6736(79)90947-4. PMID 85109
- [Background] Davies GK, Tolhurst-Cleaver CL, James TL. Respiratory depression after intrathecal narcotics. Anaesthesia. 1980 Nov;35(11):1080-3. doi: 10.1111/j.1365-2044.1980.tb05047.x. PMID 6893789
- [Background] Soni AK, Miller CG, Pratt SD, Hess PE, Oriol NE, Sarna MC. Low dose intrathecal ropivacaine with or without sufentanil provides effective analgesia and does not impair motor strength during labour: a pilot study. Can J Anaesth. 2001 Jul-Aug;48(7):677-80. doi: 10.1007/BF03016202. PMID 11495875
- [Background] Carvalho B. Respiratory depression after neuraxial opioids in the obstetric setting. Anesth Analg. 2008 Sep;107(3):956-61. doi: 10.1213/ane.0b013e318168b443. PMID 18713913
- [Background] Fuller JG, McMorland GH, Douglas MJ, Palmer L. Epidural morphine for analgesia after caesarean section: a report of 4880 patients. Can J Anaesth. 1990 Sep;37(6):636-40. doi: 10.1007/BF03006481. PMID 2208533
- [Result] Darío José PS, Ricardo N, Pedro H, Viviana C, Andrea G, Andrés G et al . Randomized double-blind controlled clinical trial for the evaluation of post-partum analgesia using epidural morphine: analgesic effectiveness of different dose regimes compared with placebo. Rev. colomb. anestesiol. 2012 Apr [cited 2021 May 04] ; 40( 1 ): 8-13. Available from: http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S0120-33472012000100004&lng=en. https://doi.org/10.1016/S0120-3347(12)70004-7.